CLINICAL TRIAL: NCT00319592
Title: Randomized, Double-blind, Phase II Study of the Safety, Tolerability and Immunogenicity Following Administration of Live Attenuated JE Vaccine (ChimeriVax™ JE) Compared With Mouse Brain-derived Inactivated JE Vaccine (JE VAX®).
Brief Title: A Safety and Efficacy Study of Two Japanese Encephalitis Vaccines ChimeriVaxTM-JE and JE-VAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-008
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Japanese Encephalitis
Keywords: Japanese encephalitis; ChimeriVax™-JE; JE-VAX®
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChimeriVax™-JE (Experimental): Subjects received 2 injections of placebo (normal saline), 1 each on Days 0 and 7, and 1 injection of ChimeriVax™-JE on Day 28.
  Interventions: Biological: ChimeriVax™-JE vaccine
- JE-VAX® (Active Comparator): Subjects received 1 injection of JE-VAX® each on Days 0, 7, and 28.
  Interventions: Biological: JE-VAX® vaccine

INTERVENTIONS:
Biological: ChimeriVax™-JE vaccine — 0.5 mL, subcutaneously
  Other Names: ChimeriVax™-JE
  Arms: ChimeriVax™-JE
Biological: JE-VAX® vaccine — 1.0 mL, subcutaneously
  Other Names: JE-VAX®
  Arms: JE-VAX®

SUMMARY:
The purpose of this study is to determine non-inferiority in seroconversion and to compare the safety and tolerability between ChimeriVax™-JE and JE-VAX® to the respective homologous virus strain and several wild types strains after completion of vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Aged ≥18 to <49 years.
* In good general health.
* Available for the study duration, including all planned follow-up visits.
* Females must have negative pregnancy test and be using adequate form of contraception

Exclusion Criteria:

* Clinically significant abnormalities on laboratory and vital sign assessments.
* Anaphylaxis or other serious adverse reactions
* Administration of another vaccine within 30 days of study treatment period.
* Physical examination indicating any significant medical condition.
* Intention to travel out of the area prior to the study visit on Day 56.
* Seropositive to Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV) or positive for Hepatitis B Surface Antigen.
* Pregnancy.
* Excessive alcohol consumption, drug abuse.
* Involvement in another clinical study within 60 days preceding the screening visit and during study treatment period.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Abdou, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- Clinical Pharamacology Center, Lenexa, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 18 May 2005 to 07 September 2005 at 1clinical center in the United States.
Pre-assignment Details: A total of 60 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- ChimeriVax™-JE After Placebo: Subjects received 2 injections of placebo (normal saline), 1 each on Days 0 and 7, and 1 injection of ChimeriVax™-JE on Day 28.
Period: Overall Study
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX® | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (8.82) | 29.2 (9.14) | 31 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Seroconverted to the Respective Homologous JE Vaccine Strain Up to 28 Days After the First Active Vaccination With Either ChimeriVax™-JE or JE-VAX® Vaccine
Description: Immunogenicity was determined by analyzing antibody response of subjects to the respective homologous JE vaccine strain using a serum dilution 50% plaque reduction neutralization test (PRNT50). Seroconversion was defined as a 4 fold increase in antibody titer of ≥ 1:10 at baseline, or an antibody titer of ≥ 1:10 for participants with a baseline antibody titer of < 1:10.
Time Frame: Day 0 (pre-vaccination) and up to Day 56 post-vaccination
Population: Seroconversion was assessed in all participants who were seronegative at baseline, received the complete vaccine regimen, and had no significant protocol deviations (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Number analyzed (Participants) | 29 | 26
Participants
  Day 14 | 0 | 7 [0 to 0]
  Day 28 | 0 | 16 [0 to 0]
  Day 42 | 18 | 24 [0 to 0]
  Day 56 | 29 | 21 [0 to 0]

2. Primary Outcome: Mean Antibody Titers of the Respective Homologous JE Vaccine Strain After the First Active Vaccination With Either JE-Vax ® or ChimeriVax™-JE
Description: Immunogenicity was determined by analyzing antibody response of subjects to the respective homologous JE vaccine strain using a serum dilution 50% plaque reduction neutralization test (PRNT50).
Time Frame: Day 0 up to Day 56 post-vaccination
Population: Antibody titers were assessed in all participants who were seronegative at baseline, received the complete vaccine regimen, and had no significant protocol deviations (Per Protocol Population).
Measure: Mean (Standard Deviation); unit: 1/dilutions
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Number analyzed (Participants) | 29 | 26
1/dilutions
  Day 0 | 5.0 (0.0) [5 to 5] | 5.0 (0.0) [5 to 5]
  Day 14 | 5.0 (0.0) [5 to 10240] | 15.2 (31.16) [5 to 160]
  Day 28 | 5.0 (0.0) | 36.5 (55.91)
  Day 42 | 599.8 (1915.35) | 184.6 (284.42)
  Day 56 | 3115.9 (4147.71) | 66.0 (133.28)

3. Primary Outcome: Number Participants That Were Seropositive to the Respective Homologous JE Vaccine Strain Before and Post-Vaccination With Either ChimeriVax™-JE or JE-VAX® Vaccine.
Description: Immunogenicity was determined by analyzing antibody response of subjects to the respective homologous JE vaccine strain using a serum dilution 50% plaque reduction neutralization test (PRNT50). Seropositive status for the ChimeriVax™-JE group was based on the ChimeriVax™-JE virus strain and positive status for the JE-VAX® group was based on the Nakayama virus strain. Participants were defined as seropositive if they had an antibody titer of ≥ 1:10. [Seropositive status can be 'Yes' or 'No']
Time Frame: Day 0 (Pre-vaccination) and up to Month 12 After First Dose
Population: Seropositive status was assessed in all participants who were seronegative at baseline, received the complete vaccine regimen, and had no significant protocol deviations (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Number analyzed (Participants) | 29 | 26
Participants
  Day 0 (N = 29, 26) | 0 | 0 [0 to 0]
  Day 56 (N = 29, 26) | 29 | 23 [0 to 0]
  Month 6 (N = 26, 24) | 24 | 7 [0 to 0]
  Month 12 (N = 26, 22) | 24 | 4 [0 to 0]

4. Primary Outcome: Mean Antibody Titers to the Respective Homologous JE Vaccine Strain Post Vaccination With Either ChimeriVax™-JE or JE-VAX®
Description: as for outcome 2
Time Frame: Day 0 (pre-vaccination) up to month 12 post-vaccination
Population: Antibody titers were assessed in all participants who were seronegative at baseline, received the complete vaccine regimen, and had no significant protocol deviations (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: 1/dilutions
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Number analyzed (Participants) | 29 | 26
1/dilutions
  Day 0 (N = 29, 26) | 5.0 (0.0) [5 to 5] | 5.0 (0.0) [5 to 5]
  Day 56 (N = 29, 26) | 3115.9 (4147.71) [40 to 10240] | 485.6 (994.74) [5 to 640]
  Month 6 (N = 26, 24) | 1727.3 (3308.16) [5 to 10240] | 44.4 (131.47) [5 to 640]
  Month 12 (N = 26, 22) | 228.1 (342.01) [5 to 1280] | 17.3 (36.24) [5 to 160]

5. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Adverse Event Following Vaccination With Either ChimeriVax™ JE or JE-VAX®
Description: Grade 3 (severe) adverse events were defined as incapacitating with inability to work or perform usual activity.
Time Frame: Day 0 up to Day 6 post-vaccination
Population: Adverse events were assessed in all participants who received at least one dose of study vaccine pr saline (Intent to Treat Population).
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Number analyzed (Participants) | 30 | 30
Participants
  Eye pain | 2 | 1
  Grade 3 Eye Pain | 0 | 0
  Photophobia | 3 | 1
  Grade 3 Photophobia | 0 | 0
  Abdominal Pain | 4 | 0
  Grade 3 Abdominal Pain | 0 | 0
  Diarrhoea | 2 | 4
  Grade 3 Diarrhoea | 0 | 0
  Nausea | 1 | 4
  Grade 3 Nausea | 0 | 0
  Vomiting | 0 | 1
  Grade 3 Vomiting | 0 | 0
  Chills | 2 | 1
  Grade 3 Chills | 0 | 0
  Fatigue | 5 | 4
  Grade 3 Fatigue | 0 | 0
  Feeling Hot | 6 | 0
  Grade 3 Feeling Hot | 0 | 0
  Injection Site Erythema | 0 | 2
  Grade 3 Injection Site Erythema | 0 | 0
  Injection Site Haemorrhage | 1 | 0
  Grade 3 Injection Site Haemorrhage | 0 | 0
  Injection Site Pain | 3 | 19
  Grade 3 Injection Site Pain | 0 | 0
  Malaise | 6 | 9
  Grade 3 Malaise | 0 | 1
  Contusion | 0 | 1
  Grade 3 Contusion | 0 | 0
  Excoriation | 1 | 0
  Grade 3 Excoriation | 0 | 0
  Limb Injury | 0 | 1
  Grade 3 Limb Injury | 0 | 0
  Body Temperature Increased | 1 | 0
  Grade 3 Body Temperature Increased | 0 | 0
  Arthralgia | 2 | 3
  Grade 3 Arthralgia | 0 | 0
  Myalgia | 4 | 6
  Grade 3 Myalgia | 0 | 0
  Disturbance in Attention | 1 | 0
  Grade 3 Disturbance in Attention | 0 | 0
  Dizziness | 0 | 1
  Grade 3 Dizziness | 0 | 1
  Headache | 13 | 9
  Grade 3 Headache | 0 | 0
  Lethargy | 4 | 7
  Grade 3 Lethargy | 0 | 1
  Somnolence | 8 | 6
  Grade 3 Somnolence | 0 | 0
  Pollakiuria | 1 | 0
  Grade 3 Pollakiuria | 0 | 0
  Dyspnoea | 1 | 3
  Grade 3 Dyspnoea | 0 | 0
  Pharyngolaryngeal Pain | 1 | 0
  Grade 3 Pharyngolaryngeal Pain | 0 | 0
  Sinus Congestion | 0 | 1
  Grade 3 Sinus Congestion | 0 | 0
  Erythema | 0 | 1
  Grade 3 Erythema | 0 | 0
  Pruritus | 1 | 0
  Grade 3 Pruritus | 0 | 0
  Rash | 1 | 0
  Grade 3 Rash | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after vaccination up to Month 12.
Arm/Group | ChimeriVax™-JE After Placebo | JE-VAX®
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 25/30 | 29/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax™-JE After Placebo (N=30) | JE-VAX® (N=30)
Eye pain (Eye disorders) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 5 (8)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 7 (8) | 5 (5)
Feeling Hot (General disorders) | 10 (11) | 0 (0)
Injection Site Erythema (General disorders) | 2 (2) | 9 (19)
Injection Site Haemorrhage (General disorders) | 2 (2) | 1 (1)
Injection Site Induration (General disorders) | 1 (1) | 2 (2)
Injection Site Pain (General disorders) | 4 (9) | 24 (70)
Injection Site Pruritus (General disorders) | 0 (0) | 2 (3)
Injection Site Swelling (General disorders) | 0 (0) | 6 (8)
Malaise (General disorders) | 9 (10) | 11 (11)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 3 (4)
Sunburn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
White Blood Cell Count Increased (Investigations) | 2 (2) | 2 (3)
White Blood Cells Urine Positive (Investigations) | 4 (4) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (8)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 17 (28) | 12 (25)
Lethargy (Nervous system disorders) | 5 (8) | 8 (10)
Somnolence (Nervous system disorders) | 9 (11) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.